CLINICAL TRIAL: NCT00223639
Title: New Medications to Treat Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bankole Johnson (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Bankole Johnson, Chair of Psychiatry and Neurobehavioral Sciences, University of Virginia
Organization: University of Virginia (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 5R01AA014628-02 (NIH); 5R01AA014628-02 (NIH)
Record Dates: First submitted 2005-09-19; First posted 2005-09-22 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Alcoholism
Keywords: alcoholism /alcohol abuse; alcoholism antagonist; anticonvulsant; cognition; neuropharmacology; substance abuse related behavior; craving; euphoria; relapse /recurrence; patient oriented research
MeSH Terms: conditions — Alcoholism; Recurrence | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Topiramate (Experimental)
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator)
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — 200mg twice a day
  Other Names: Topamax

SUMMARY:
In the last decade, there has been an explosion of new knowledge of the neuroscientific basis of alcohol-seeking behavior. Briefly, medications that modulate mesolimbic dopamine pathways by facilitating gamma amino butyric function and inhibiting the action of excitatory amino acids should reliably diminish alcohol's rewarding effects. Topiramate (a sulfamate-substituted fructo-pyranose derivative) has these characteristics. In support of this concept, we have shown in a phase-II-type medications clinical trial that topiramate is significantly superior to placebo at improving drinking outcomes and decreasing craving among (N = 150) alcohol-dependent individuals. Using the carefully controlled environment of the human laboratory, we are submitting a revised application containing a set of systematic studies to assess directly the mechanistic neuropharmacological processes that are associated with topiramate's anti-drinking effects. This will provide a more comprehensive understanding of the neurobiology of alcohol-seeking behavior and aid in the development of even more effective compounds for the treatment of alcohol dependence. Thus, the specific aims of the project are to: 1) determine the dose-relationship of acute effects of topiramate to reduce alcohol effects related to its abuse and addiction potential. We hypothesize that topiramate will reduce alcohol-induced craving, reward, and euphoria; 2) determine whether chronic treatment with an acutely effective dose of topiramate produces substantial reductions in alcohol-related cue-induced craving, thereby decreasing the potential for treatment relapse. We hypothesize that chronic topiramate administration will desensitize (reduce) alcohol craving produced by alcohol-related sensory cues; and 3) determine whether topiramate interactions with and without alcohol are associated with neurocognitive impairment. Clinical studies including ours have suggested that topiramate use may be associated with neurocognitive effects such as loss of concentration and memory impairment. In our own study, these effects were mild and not associated with reduced treatment compliance. Since alcohol's ability to produce neurocognitive impairment may be mediated through similar ionic mechanisms to that of topiramate, the proposed human laboratory setting affords us the unique opportunity to more clearly delineate topiramate's neurocognitive effects in both the presence and absence of alcohol. This study supports NIAAA's goal to develop effective medications for treating alcoholism and to understand the basic underpinnings of the disease.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV-R diagnosis of alcohol dependence.
* Drinking on average ≥14 and ≥21 drinks/week in the 30 days prior to enrollment for women and men, respectively, and describing a liking for and frequent use of beer as the alcohol-containing beverage.
* Good physical health as determined by a complete physical examination, electrocardiogram within normal limits, and laboratory screening tests within acceptable range (see exclusion criteria).
* Negative pregnancy test at intake. Women of childbearing potential will be placed on oral contraceptives and also will be expected to use barrier and spermicide as an additional form of contraception if sexually active.
* Literate in English language, and able to read, understand, and complete rating scales and questionnaires accurately.
* Willingness to comply with study procedures and protocol including agreement to overnight stay at the human laboratory. Compliance with the alcohol, tobacco, and drug-free environment regulations at the human laboratory is also a condition of enrollment.
* Written informed consent.

Exclusion Criteria:

* Expression of desire for immediate treatment for alcohol or drug addiction.
* History of mental illness that warrants treatment or would preclude safe participation in the protocol except nicotine dependence, as determined by mental status and psychiatric interview using the Structured Clinical Interview for DSM-IV.
* Acute or chronic organic brain syndrome, schizophrenia, bipolar disorder, or any psychotic disorder.
* Significant medical illness (including hypertension) as determined by history and/or complete physical examination.
* Uncontrolled uterine or cervical bleeding.
* History of blood clots.
* Past problems with oral contraceptive pills.
* Gross neurological disease.
* Mental retardation.
* Neurocognitive functioning >1.5 standard deviation below expected range
* Clinically significant abnormalities on the electrocardiogram that will preclude safe participation.
* History of ischemic heart disease or myocardial infarction.
* History of glaucoma or thyroid disease.
* Current infective hepatitis as evidenced by clinical manifestations..
* Positive pregnancy test.
* Women 35 and above who smoke will be excluded from participating in this research study.
* Participation in a human laboratory or clinical study within the last 30 days.
* Clinically significant laboratory screening test (LST) results on hematology, chemistry, or urine analysis as defined by the FDA Neuropharmacology Division guidelines. Elevation of liver enzymes (SGOT), serum glutamic pyruvic transaminase (SGPT), blood urea nitrogen (BUN), or lactate dehydrogenase (LDH) - up to ×4 above the normal range - will be allowed unless there is evidence of hepatocellular disease or failure. In addition, we will test for hematocrit as more than 300 ml of blood will be taken during study 1. Hematocrit levels must be > 41% for males and > 38% for females.
* For study 1, persons weighing less than 110 lbs will be excluded, due to the amount of blood taken in study 1 (more than 300 ml).
* History of any severe or life-threatening reaction to topiramate
* Past or current history of seizures.
* Past or current history of kidney stones.
* Use of any carbonic anhydrase medication.
* Being treated with any medication with potential interactions with alcohol or topiramate.
* Pending imprisonment.
* For smokers, previous adverse reaction to nicotine patch.
* Reporting no experience of craving for alcohol (by self-report).
* Postmenopausal women will not be recruited into this study.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2005-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Reduction of alcohol-induced craving,reward,and euphoria | During testing days

SECONDARY OUTCOMES:
Reductions in alcohol-related cue-induced associated with relapse | During testing days
Determine whether topiramate interactions with and without alcohol are associated with neurocognitive impairment | During testing days

CONTACTS AND LOCATIONS:
Overall Officials: Bankole A Johnson, DSc,MD,PhD, Principal Investigator — University of Virginia
Locations (2):
- United States (2):
  - UVA CARE, Charlottesville, Virginia
  - UVA CARE Richmond, Richmond, Virginia